CLINICAL TRIAL: NCT00740415
Title: First-line Treatment of Mantle Cell Lymphoma of Old Patients . Evaluate the Efficacy, Toxicity, and Molecular Prognostic Factors of Velcade®) in Association With Chemotherapy and Immunotherapy With Rituximab
Brief Title: Rituximab, Bortezomib,Bendamustine , Dexamethasone, Patients With Mantle Cell Lymphoma
Acronym: ManteauRiBVD
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: French Innovative Leukemia Organisation (Other)
Collaborators: Janssen, LP (Industry); Mundipharma Pte Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000589544; -MANTEAU-2010-SA (Other: FILO)
Record Dates: First submitted 2008-08-22; First posted 2008-08-25 (Estimated); Last update posted 2016-03-16 (Estimated); Status verified 2016-03

CONDITIONS: Lymphoma
Keywords: contiguous stage II mantle cell lymphoma; noncontiguous stage II mantle cell lymphoma; stage III mantle cell lymphoma; stage IV mantle cell lymphoma
MeSH Terms: conditions — Lymphoma; Lymphoma, Mantle-Cell | interventions — Rituximab; Bortezomib; Dexamethasone; Bendamustine Hydrochloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- ARM RiBVD (Experimental): RiBVD 6 cycles every 28 days day 1 :
  * Rituximab /Mabthera®, 375 mg/m2 en IV
  * Bendamustine, 90 mg/m2 en IVD
  * Bortezomib/Velcade®, 1,3 mg/m2 en IVD day 2 : - Bendamustine, 90 mg/m2 en IVD
  * Dexamethasone, 40 mg IV day 4 : - Bortezomib/Velcade®, 1,3 mg/m2 en IVD day 8 : - Bortezomib/Velcade®, 1,3 mg/m2 en IVD day 11 : - Bortezomib/Velcade®, 1,3 mg/m2 en IVD
  Interventions: Biological: rituximab; Drug: bortezomib; Drug: dexamethasone; Drug: Bendamustine

INTERVENTIONS:
Biological: rituximab — Rituximab, 375 mg/m2 Intraveinous
  Other Names: Mabthera ®,
Drug: bortezomib — -Velcade®, 1,3 mg/m2 Intraveinous on days 1, 4, 8 and 11
  Other Names: Velcade
Drug: dexamethasone — day - Dexamethasone, 40 mg Intraveinous
Drug: Bendamustine — -Day 1 and day 2 Bendamustine/Levact ®,, 90 mg/m2 Intraveinous
  Other Names: Levact ®

SUMMARY:
RATIONALE: Monoclonal antibodies, such as rituximab, can block cancer growth in different ways. Some block the ability of cancer cells to grow and spread. Others find cancer cells and help kill them or carry cancer-killing substances to them. Bortezomib may stop the growth of cancer cells by blocking some of the enzymes needed for cell growth and by blocking blood flow to the tumor. Drugs used in chemotherapy, such as doxorubicin, dexamethasone, and chlorambucil, work in different ways to stop the growth of cancer cells, either by killing the cells or by stopping them from dividing. Giving combination chemotherapy together with rituximab and bortezomib may kill more cancer cells.

PURPOSE: This phase II trial is studying how well giving rituximab together with bortezomib, doxorubicin, dexamethasone, and chlorambucil works as first-line therapy in treating older patients with stage II, stage III, or stage IV mantle cell lymphoma.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Evaluate the efficacy of rituximab, bortezomib, doxorubicin hydrochloride, dexamethasone, and chlorambucil as first-line therapy in patients with stage II-IV mantle cell lymphoma.

Secondary

* Determine the complete response rate in these patients.
* Determine the efficacy, in terms of complete and overall response, by F18 fludeoxyglucose scan.
* Determine overall, disease-free, and event-free survival of these patients.
* Assess tolerability of this regimen in these patients.
* Evaluate the impact of factors, described in previous protocols, on response to therapy and survival.
* Assess the impact of residual disease in cerebrospinal fluid on survival.

OUTLINE: This is a multicenter study.

Patients receive rituximab IV on day 1 (days 1 and 8 of the first course only); bortezomib IV on days 1, 4, 8, and 11; doxorubicin hydrochloride IV continuously over 24 hours on days 1-4; dexamethasone IV on days 1-4; and oral chlorambucil on days 20-29. Treatment repeats every 5 weeks for 4 courses in the absence of disease progression or unacceptable toxicity.

Patients who achieve at least 50% response receive 2 additional courses of therapy.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of mantle cell lymphoma

  * Stage II-IV disease
* No neuromeningeal disease

PATIENT CHARACTERISTICS:

* WHO performance status 0-2
* No prior cancer except for carcinoma in situ of the cervix or basal cell skin cancer
* LVEF > 50%
* HIV-negative
* Hepatitis B- and C-negative
* No hepatocellular, renal, or bone marrow insufficiency unrelated to lymphoma

PRIOR CONCURRENT THERAPY:

* Not specified

Ages: 65 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 39 (Actual)
Dates: Start 2007-06; Primary Completion 2011-05 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
Overall response rate after 4 courses of therapy | 4 months

CONTACTS AND LOCATIONS:
Overall Officials: Remy Gressin, MD, Study Chair — CHU de Grenoble - Hopital de la Tronche
Locations (1):
- CHU de Grenoble - Hopital Michallon, Grenoble, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: FILO website — http://www.filo-leucemie.org